CLINICAL TRIAL: NCT02721745
Title: Cause and Consequence of Neural Fatigue
Acronym: Fatstim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C15-59; 2015-A01445-44 (Registry Identifier: IRDB)
Record Dates: First submitted 2016-03-03; First posted 2016-03-29 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Fatigue
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Natural Fatigue (Experimental): Brain activity will be record through EEG (physiological measure),O2 consumption will be record through a metabolic monitor (physiological measure), or eye tracker according to the group.
  Interventions: Behavioral: Natural Fatigue
- tDCS anodal (Experimental): Brain activity will be record through EEG (physiological measure),O2 consumption will be record through a metabolic monitor (physiological measure), or eye tracker according to the group.
  Interventions: Device: tDCS
- tDCS cathodal (Experimental): Brain activity will be record through EEG (physiological measure),O2 consumption will be record through a metabolic monitor (physiological measure), or eye tracker according to the group.
  Interventions: Device: tDCS
- tDCS sham (Experimental): Brain activity will be record through EEG (physiological measure),O2 consumption will be record through a metabolic monitor (physiological measure), or eye tracker according to the group.
  Interventions: Device: tDCS
- inhibitory TMS (Experimental): Brain activity will be record through EEG (physiological measure),O2 consumption will be record through a metabolic monitor (physiological measure), or eye tracker according to the group.
  Interventions: Device: TMS
- Sham TMS (Experimental): Brain activity will be record through EEG (physiological measure),O2 consumption will be record through a metabolic monitor (physiological measure), or eye tracker according to the group.
  Interventions: Device: TMS

INTERVENTIONS:
Behavioral: Natural Fatigue — Experimental: EEG Indirect Calorimetry Pupillometry
  Arms: Natural Fatigue
Device: tDCS — Experimental: EEG Indirect Calorimetry Pupillometry
  Arms: tDCS anodal; tDCS cathodal; tDCS sham
Device: TMS — Experimental: EEG Indirect Calorimetry Pupillometry
  Arms: Sham TMS; inhibitory TMS

SUMMARY:
While the scientific community understands quite well why muscles ache after prolonged exercise, the origins of mental fatigue remain totally mysterious. Existing theories remain at a psychological level, with scarce supporting evidence. Mental fatigue typically occurs after long episodes during which humans exert control on motor or cognitive processes, instead of executing routine or stimulus-driven behaviours. However, work organization (especially in risky job like airplane control or medical profession) and pathologies due to an overload of work (like burn-out) seems to be directly linked to neural fatigue. One of the consequences of neural fatigue is to alter decision-making. As an example, the choice between an immediate monetary reward and a larger but delayed monetary reward (the so called intertemporal choices) are susceptible to fatigue state of its underpinning neural network.

The investigators are proposing an exploratory study of neural fatigue, induced either in a natural way (by performing cognitive tasks for hours) or by transcranial stimulation, using three main physiological measures (Electro-encephalography to measure neural activity, indirect calorimetry to measure the metabolic cost of a cognitive effort, and pupillometry to measure cognitive effort).

This study should allow to better understand the consequences of neural fatigue on cognitive functions like decision making as well as the associated physiological variables.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed people;
* between 20 à 39 years old;
* able to understand the instructions and to perform the behavioral tasks of the study ;
* informed consent to take part to the study (signature of a a consent form);
* people being registered to social security or universal medical protection or equivalent;

Exclusion Criteria:

For each experiment:

* neurological, psychiatric or serious illness history
* ongoing or recently stopped (lower than three weeks) psychotropic treatment;
* excessive psychotropic substances consumption or chronical consumption the examination day;
* People being not able to perform the tasks (alteration of one of the cognitive functions or elementary visual disorder avoiding the identification of the experimental stimuli);
* adult under legal protection (guardianship, or under the protection of a conservator);
* adult people being not able to express his consent;
* people being deprived of liberty as a consequence of an administrative or judicial decision;
* pregnant, parturient or nursing women;
* people taking part to another biomedical study or still being in the exclusion phase of another research;
* hospitalized people without consent;
* people who could not participate to the full study for any reasons.

For the experiments involving transcranial stimulation, in addition to the previous ones:

* take of drugs known to lower the epileptogenic threshold;
* take of barbiturate, gabapentin, topiramate, clonazepam in the 7 days before the first visit;
* history of awareness loss;
* people having contraindication for having a transcranial magnetic stimulation or for having an MRI examination;
* People who does not want to be informed of any significant irregularity that could be detected during the MRI examination;
* claustrophobic people ;

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Proportion of chosen immediate reward in intertemporal questions between an immediate reward smaller than a delayed reward. | Day 0
  Several questions between two options (an immediate reward and and a larger delayed reward) will be asked to the participants through a computer. The measure of impulsivity corresponds to the proportion of immediate reward that wil be chosen through the keyboard (left or right arrows).
Physiological Measures: EEG | Day 0
  power of electrical brain oscillation.
Physiological Measures: indirect calorimetry | day 0
  volume of O2 consumption and CO2 expulsion.
Physiological Measures:pupillometry | Day 0
  pupil dilation.

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, Paris, France

IPD SHARING:
Plan to Share IPD: No